CLINICAL TRIAL: NCT06613880
Title: A Prospective, Single Center, Single-arm Study on the Efficacy and Safety of Standard Immunosuppressive Therapy Combined With Romiplostim N01 as First-line Treatment for Severe Aplastic Anemia
Brief Title: Standard Immunosuppressive Therapy Combined With Romiplostim N01 as First-line Treatment for Severe Aplastic Anemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024070
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-09

CONDITIONS: Aplastic Anemia; TPO Receptor Agonists
Keywords: Severe aplastic anemia; Romiplostim N01
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- p-ALG+Romiplostim N01+CsA (Experimental): The maximum screening period was 4 weeks, and after entering the treatment period, the patients were treated with p-ALG combined with cyclosporine and Romiplostim N01. Symptomatic leukocyte elevation, blood transfusion support, and anti-infective therapy are allowed during this period, according to the patient's blood routine. If a patient has a serious adverse event during treatment, it will be treated according to the criteria for suspension and recovery.
  Interventions: Drug: standard IST combined with Romiplostim N01

INTERVENTIONS:
Drug: standard IST combined with Romiplostim N01 — Romiplostim N01 is a class of TPO receptor agonists. Its TPO peptide can bind to TPO receptors on megakaryocyte precursors in the bone marrow and activate them, triggering a series of intracellular signalling pathways, including JAK2/STAT5, PI3K/Akt, MEK/ERK, and p38, which ultimately lead to gene transcription and increased megakaryocyte proliferation and differentiation.

SUMMARY:
This prospective, single center, single-arm study aims to evaluate the efficacy and safety of anti-human T lymphocyte porcine immunoglobulin (p-ALG) in combination with cyclosporine and Romiplostim in treating severe aplastic anemia (SAA). It will include 48 patients with newly diagnosed SAA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years
* Diagnosis of severe or very severe aplastic anemia
* Patients are unconditionally or unacceptable undergoing allogeneic hematopoietic stem cell transplantation
* ECOG performance status ≤2
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* Received > 4 weeks of TPO-RA drug before treatment
* Received > 4 weeks of immunosuppressive therapy before treatment
* History of thromboembolic disease
* Intolerance to Romiplostim N01 or cyclosporine
* Allergy to ALG
* Presence of uncontrolled active infection
* Presence of uncontrolled hypertension (≥140/90mmHg), diabetes mellitus (fasting blood glucose≥ 7.0 mmol/L or random blood glucose ≥ 11.1 mmol/L)
* Abnormal liver and kidney function: Aspartate Transaminase (AST) or Alanine Transaminase (ALT) > 3 ULN, creatinine ≥ 2.5 ULN
* History of chemoradiotherapy for malignant solid tumors
* History of other systemic serious illnesses
* Females who are pregnant/lactating or need pregnancy
* Patients considered to be ineligible for the study by the investigator for reasons other than the above

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Within 27 weeks post treatment
  Percentage of patients with hematological response, including complete response (CR) or partial response (PR). Hematological response is evaluated by hemoglobin (Hb), platelet count (PLT) and absolute neutrophil count (ANC).

SECONDARY OUTCOMES:
Overall response rate | Within 3 months post treatment
  Percentage of patients with hematological response, including complete response (CR) or partial response (PR). Hematological response is evaluated by hemoglobin (Hb), platelet count (PLT) and absolute neutrophil count (ANC).
Time to hematological response | Within 27 weeks post treatment
  Duration time was calculated from enrollment to achieve hematological response.
Incidence of adverse events | Within 27 weeks post treatment
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Regenerative Medicine Center and Red Blood Cell Disorders Center, Tianjin, Tianjin Municipality, China